CLINICAL TRIAL: NCT05417750
Title: An Open-label, Single-arm, Phase I Study to Evaluate the Safety and Efficacy of Autologous Tumor Infiltrating Lymphocytes Injection in Patients With Advanced Malignant Solid Tumors
Brief Title: A Phase I Study of GC101 TIL in Advanced Solid Tumors
Acronym: MIZAR-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Juncell Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GC101 TIL-ST-01
Record Dates: First submitted 2022-05-31; First posted 2022-06-14 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Tumor Infiltrating Lymphocytes; Safety; Advanced Solid Tumor; Immunotherapy; Efficacy; Adverse Drug Event
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Experimental: Cohort 1 (Experimental): dose escalation group: participants with advanced solid tumors using cryopreserved GC101 TIL
  Interventions: Drug: TIL therapy
- Experimental: Cohort 2 (Experimental): participants with advanced malignant melanoma using cryopreserved GC101 TIL
  Interventions: Drug: TIL therapy
- Experimental: Cohort 3 (Experimental): participants with advanced NSCLC using cryopreserved GC101 TIL
  Interventions: Drug: TIL therapy
- Experimental: Cohort 4 (Experimental): participants with advanced HNSCC using cryopreserved GC101 TIL
  Interventions: Drug: TIL therapy
- Experimental: Cohort 5 (Experimental): participants with advanced cervical cancer using cryopreserved GC101 TIL
  Interventions: Drug: TIL therapy

INTERVENTIONS:
Drug: TIL therapy — A tumor sample is resected from each participant and cultured ex vivo to expand the population of autologous tumor infiltrating lymphocytes injection (GC101 TIL). After lymphodepletion, patients are infused GC101 TIL followed sintilimab.

SUMMARY:
20-60 participants are expected to be enrolled for the Phase I clinical trial which is further divided into two parts: a "3+3" dose escalation study and an expanded enrollment study.

The Phase I clinical trial is expected to be finished in 36 months. To be specific, the dose escalation study plans to include patients with advanced malignant solid tumors with clear pathological diagnosis, including melanoma, cervical cancer, head and neck squamous cell tumors, non-small cell lung cancer and breast cancer, etc.; while the expanded enrollment study plans to include those with melanoma, cervical cancer, and head and neck squamous cell tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be ≥18 and ≤75 years of age at the time of consent.
2. Patients with advanced metastatic solid tumors with clear pathological diagnosis, including melanoma, cervical cancer, head and neck squamous cell tumors, non-small cell lung cancer and breast cancer, etc.; while the expanded enrollment study plans to include those with melanoma, cervical cancer, and head and neck squamous cell tumors.
3. At least one measurable target lesion even after resection, as defined by RECIST1.1.

   Lesions in previously irradiated areas (or other local therapy) should not be selected as target lesions, unless treatments was ≥3 months prior to Screening, and there has been demonstrated disease progression in that particular lesion.
4. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Patients must have an estimated life expectancy of ≥3 months.
6. In the opinion of the Investigator, patients must be able to sign the ICF and complete all study-required procedures.
7. Patients must have the following hematologic parameters, Coagulation functions and hepatic and renal function:

   * White Blood Cell (WBC)≥2.5×10^9/L；
   * Absolute Lymphocyte Count (ANC)≥1.5×10^9/L;
   * Absolute Lymphocyte Count(ALC)≥0.7×10^9/L;
   * Platelet≥100×10^9/L；
   * International Normalized Ratio（INR）≤1.5×ULN;
   * Activated Partial Thromboplastin Time（APTT）≤1.5×ULN;
   * Serum Creatinine (Scr)≤1.5mg/dL (or 132.6μmol/L) or Creatinine Clearance≥60mL/min
   * Urinalysis: urine protein less than 2+, or 24-hour urine protein <1g;
   * Alanine aminotransferase(AST/SGOT) ≤3×ULN;
   * Alanine aminotransferase (ALT/SGPT) ≤3×ULN;
   * Total Bilirubin(TBIL)≤1.5×ULN；
8. Patients must have a washout period ≥ 4 weeks from prior anticancer therapy(ies) to the start of the planned preconditioning regimen, including targeted therapy, chemotherapy, immunotherapy: anti-cytotoxic T lymphocyte-associated antigen 4 (CTLA-4)/anti-PD-1, other monoclonal antibody (mAb), or vaccine Palliative radiation therapy.
9. Patients of childbearing potential or their partners of childbearing potential must be willing to take the appropriate precaution to avoid pregnancy or fathering a child for the duration of the study and practice an approved, highly effective method of birth control during treatment and for 12 months after receiving the last protocol-related therapy.
10. Patients must have no contraindications for surgery or biopsy.
11. Patients (or legally authorized representative) must have the ability to understand the requirements of the study, have provided written informed consent as evidenced by signature on an ICF approved by an Institutional Review Board/Independent Ethics Committee (IRB/IEC), and agree to abide by the study restrictions and return to the site for the required assessments, including the OS Follow-up Period.

Exclusion Criteria:

1. Patients have not recovered from all prior therapy-related adverse events (AEs) to ≤ Grade 1 (per Common Terminology Criteria for Adverse Events [CTCAE] v5.0), except for alopecia or vitiligo, prior to Enrollment (tumor resection).
2. Patients who have received an organ allograft or prior cell transfer therapy.
3. Patients with symptomatic and/or untreated brain metastases (of any size and any number).
4. Patients who are on chronic systemic steroid therapy for any reason.
5. Patients who have active medical illness(es) that would pose increased risk for study participation, including: active systemic infections requiring systemic ABX, coagulation disorders, or other active major medical illnesses of the cardiovascular, respiratory, or immune system.
6. Patients with systemic active infection requiring treatment, with positive blood culture or imaging evidence of infection, including active tuberculosis.
7. Patients with hepatic encephalopathy, hepatorenal syndrome, Child-Pugh class B or more severe cirrhosis, or liver failure.
8. Uncontrolled arterial hypertension（SBP≥160mmHg and/or DBP≥100mmHg）or any unstable cardiovascular or cerebrovascular disease in the recent 6 months of consent.
9. Patients who have a left ventricular ejection fraction (LVEF) < 50% or New York Heart Association (NYHA) functional classification Class 3 or Class 4.
10. Female patients who are pregnant or breastfeeding.
11. Patients who are HIV positive, positive syphilis serological test, positive COVID-19 nucleic acid test, or clinically active hepatitis A, B, and C including virus carriers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Maximal Tolerance Dose | Up to Day 28
Dose Limiting Toxicity | Up to Day 28
Adverse Events | Maximum 360 days

SECONDARY OUTCOMES:
Disease Assessment for Duration of Response | Every 6 weeks for 12 months
  Evaluate the efficacy endpoints of DOR by the investigator with RECIST v1.1 and iRECIST
Disease Assessment for Disease Control Rate | Every 6 weeks for 12 months
  Evaluate the efficacy endpoints of DCR by the investigator with RECIST v1.1 and iRECIST
Disease Assessment for Progression-Free Survival | Every 6 weeks for 12 months
  Evaluate the efficacy endpoints of PFS by the investigator with RECIST v1.1 and iRECIST
Disease Assessment for Objective Response Rate | Every 6 weeks for 12 months
  Evaluate the efficacy endpoints of ORR by the investigator with RECIST v1.1 and iRECIST
Quality of Life Assessment | Every 6 weeks for 12 months
  Evaluate with EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No